CLINICAL TRIAL: NCT03058965
Title: Phase 0 Evaluation of [18F]MNI-958 as a Potential PET Radioligand for Imaging Tau Protein in the Brain of Patients With Probable Alzheimer's Disease or Progressive Supranuclear Palsy Compared With Healthy Volunteers
Brief Title: Phase 0 Evaluation of [18F]MNI-958 as a Potential PET Radioligand for Imaging Tau Protein in the Brain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-958
Record Dates: First submitted 2017-01-12; First posted 2017-02-23 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer Disease; Healthy Volunteers; Progressive Supranuclear Palsy
Keywords: AD; HV; PSP
MeSH Terms: conditions — Alzheimer Disease; Supranuclear Palsy, Progressive | interventions — florbetapir; ioflupane

ARMS (1):
- [18F]MNI-958 (Experimental): To evaluate [18F]MNI-958, a tau targeted PET radioligand.
  Interventions: Drug: [18F]MNI-958; Drug: [18F]Florbetapir; Drug: DaTscan

INTERVENTIONS:
Drug: [18F]MNI-958 — Subjects will undergo PET imaging using [18F]MNI-958, a PET radioligand for imaging tau.
Drug: [18F]Florbetapir — Subjects with Alzheimer's disease will receive a [18F]florbetapir scan to compare distribution of tau in the brain compared to that of [18F]MNI-958.
Drug: DaTscan — DaTscan SPECT imaging will be completed in those PSP subjects who have not previously had DATScan imaging as part of the screening procedures.

SUMMARY:
The overall goal of this imaging trial is to evaluate [18F]MNI-958, a tau targeted PET radioligand, in individuals with Alzheimer's disease (AD), Progressive Supranuclear Palsy (PSP), and healthy volunteers (HV).

ELIGIBILITY:
Inclusion:

* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to use a barrier contraception method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
* Male subjects must not donate sperm for the study duration.
* Willing and able to cooperate with study procedures

Inclusion Criteria for Healthy Volunteer Subjects:

* Males and females aged ≥50 years. Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]MNI-958 imaging visit.
* No cognitive impairment from neuropsychological battery as judged by the investigator
* Have screening [18F]florbetapir PET imaging demonstrating no significant amyloid binding based on qualitative analysis (visual read).
* No family history of Alzheimer's disease or neurological disease associated with dementia
* Have a CDR score=0

Inclusion Criteria for subjects with a diagnosis of probable Alzheimer's disease (AD):

* Males and females aged 50 to 90 years.
* Have probable Alzheimer's disease, based on the NINCDS/ADRDA and DSM-IV criteria.
* Have a CDR score of 0.5 or greater at screening.
* Have an MMSE score ≤ 28.
* Have screening or prior (in the last 12 months) [18F]florbetapir PET imaging demonstrating amyloid binding based on qualitative (visual read)
* A brain MRI that supports a diagnosis of AD, with no evidence of focal disease to account for dementia or MRI exclusion criteria.
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 30 days before the screening visit.
* Signed and dated written informed consent obtained from the subject and the subject's legally authorized representative or caregiver (if applicable).
* The subject has an appropriate caregiver capable of accompanying subject, if necessary.

Inclusion Criteria for subjects with a diagnosis of probable Progressive Suprnuclear Palsy (PSP)

* Males and females aged 50 to 90 years.
* Has a clinical diagnosis of PSP based on the NINDS and Society for PSP criteria (Litvan, et al 1996).
* Have screening or prior DaTscan SPECT imaging demonstrating evidence of dopamine transporter deficit based on visual read.
* A brain MRI that supports a diagnosis of PSP, with no other evidence of significant neurologic pathology
* Medications taken for symptomatic treatment of PSP must be maintained on a stable dosage regimen for at least 30 days before screening visit.
* Signed and dated written informed consent obtained from the subject and the subject's legally authorized representative or caregiver (if applicable).
* The subject has an appropriate caregiver capable of accompanying subject, if necessary.

Exclusion Criteria:

* Current or prior history of any alcohol or drug abuse.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Subject has received an investigational drug or device within 30 days of screening
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines
* Pregnancy, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* MRI exclusion criteria include: evidence of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the FLAIR sequence that is ≥20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with CNS disease.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.

Exclusion Criteria for Subjects with Probable AD:

* Has received treatment that targeted amyloid-β or tau within the last 3 months.

Exclusion Criteria for Subjects with Probable PSP:

* Ongoing treatment with methylphenidate, bupropion, modafinil, metoclopramide, alpha methyldopa, reserpine, or amphetamine derivative.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Tracer uptake will be evaluated in regions of interest for analysis of regional [18F]MNI-958 binding/uptake and expressed in SUV by using established methods for normalization for 3 AD, 3 PSP, and 3 HV subjects. | 1 year
  Descriptive statistics will be applied to describe the tau deposition by region as measured by [18F]MNI-958.

CONTACTS AND LOCATIONS:
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — https://mnimaging.com/